CLINICAL TRIAL: NCT06141941
Title: Does the Use of Continuous Glucose Monitoring (CGM) in the Immediate Postpartum Period in Women With Pregestational Diabetes Admitted to the Hospital Decrease Hypoglycemic Episodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea L. Greiner (Other)
Responsible Party: Sponsor-Investigator, Andrea L. Greiner, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202101006
Record Dates: First submitted 2023-10-23; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pregestational Diabetes
Keywords: postpartum; type 1 diabetes; type 2 diabetes; continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CGM (Other): A CGM device (Dexcom sensor and transmitter) will be placed by research personnel upon presentation to Labor and Delivery unit.
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Continuous glucose monitoring

SUMMARY:
This study will examine whether continuous glucose monitoring in patients hospitalized in the immediate postpartum period is more effective than traditional point of care glucose testing in identifying patients with hypoglycemia.

DETAILED DESCRIPTION:
This is a prospective cohort study of women with type 1 and type 2 diabetes in the postpartum period. After obtaining informed consent, a CGM device (Dexcom sensor and transmitter) will be placed by research personnel upon presentation to labor or in prenatal clinic if seen within 3 days of planned induction of labor or planned cesarean section. Patient will be assisted in getting the Dexcom G6 app on their cell phone to be the receiver of glucose data. Patients who are currently using the Dexcom CGM for routine monitoring of their glucoses, will be allowed to continue using their own sensor and transmitter. Upon presentation to Labor and Delivery, patients will be assisted in activating the Share App on their cell phone. Labor and Delivery Nursing Staff will be given a Samsun phone with the Follow app in order to receive glucose data. The Samsung phone will be transferred to the Mother/Baby Unit with the patient after delivery.

Glucose values from the CGM device will then be available to nursing through the Samsung phone. Nursing will be able to see current glucose data on their patient and would receive alarms to indicate hypoglycemia or impending hypoglycemia. Nursing will be provided with instructions for how to access the CGM follow app and how to appropriately respond to the alarms. Nursing will continue to perform standard of care blood glucose monitoring per routine protocol but will also obtain a finger stick to validate a blood glucose level whenever a low CGM alarm sounds. Low blood glucose values <70 mg/dl will be treated per local institutional nursing policy. Monitoring of glucose levels through the CGM device will continue throughout their postpartum hospital stay. This is typically 2 days for a vaginal delivery, 3 days for a cesarean section. Patients who do not use CGM as part of their routine care, will have their CGM sensor and transmitter removed prior to discharge from the hospital.

Following discharge from the hospital, there will be no additional long term follow-up.

Data we plan to collect for analysis includes: type of diabetes (DM1/DM2), point of care glucose values, number of hypoglycemic events, number of times treated for hypoglycemia.

ELIGIBILITY:
Inclusion:

1- Individuals in the third trimester of pregnancy admitted to the hospital with diabetes type 1 or diabetes type 2, own a smart device (which will serve as a receiver for the CGM device)

Exclusion:

1. Patients less than 18 years of age
2. non-English speaking patients
3. gestational diabetes
4. extensive skin changes/diseases that inhibit wearing a sensor on normal skin, known allergy to adhesives

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Glucose values | Postpartum admission, 2-4 days
  glucose values obtained from CGM application

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Greiner, MD, Principal Investigator — University of Iowa OBGYN
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Background] Spanakis EK, Levitt DL, Siddiqui T, Singh LG, Pinault L, Sorkin J, Umpierrez GE, Fink JC. The Effect of Continuous Glucose Monitoring in Preventing Inpatient Hypoglycemia in General Wards: The Glucose Telemetry System. J Diabetes Sci Technol. 2018 Jan;12(1):20-25. doi: 10.1177/1932296817748964. Epub 2017 Dec 13. PMID 29237288
- [Background] Singh LG, Satyarengga M, Marcano I, Scott WH, Pinault LF, Feng Z, Sorkin JD, Umpierrez GE, Spanakis EK. Reducing Inpatient Hypoglycemia in the General Wards Using Real-time Continuous Glucose Monitoring: The Glucose Telemetry System, a Randomized Clinical Trial. Diabetes Care. 2020 Nov;43(11):2736-2743. doi: 10.2337/dc20-0840. Epub 2020 Aug 5. PMID 32759361